CLINICAL TRIAL: NCT06116136
Title: Open Label, Non-randomized, Phase 1b/2 Trial Investigating the Safety, Tolerability, and Antitumor Activity of S095029 (Anti-NKG2A Antibody) as a Part of Combination Therapy in Participants With Locally Advanced and Unresectable or Metastatic MSI-H/dMMR Gastro-esophageal Junction /Gastric Cancer
Brief Title: A Study to Evaluate the Safety and the Activity of S095029 as Part of Combination Therapy in Advanced Gastroesophageal Junction/Gastric Cancers.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95029-002; Keynote E70 (Other: Merck); 2023-507995-33 (EudraCT Number); MK-3475-E70 (Other: Merck)
Record Dates: First submitted 2023-09-28; First posted 2023-11-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: MSI-H/dMMR Gastroesophageal-junction Cancer; MSI-H/dMMR Gastric Cancer
Keywords: Anti-NKG2A; S095029; pembrolizumab; MSI-H/dMMR; Gastric cancer; Gastroesophageal-junction cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S095029 and pembrolizumab (Experimental): Participants diagnosed with gastric cancer (GC) or gastroesophageal junction cancer (GEJ), not previously treated with checkpoint inhibitors (CPIs) may first be enrolled into a Phase 1b safety lead-in part which will be used to identify the recommended Phase 2 dose (RP2D) of S095029 in combination with pembrolizumab. During the Phase 2 part, participants will receive the recommended Phase 2 dose (RP2D) of S095029, along with pembrolizumab.
  Interventions: Drug: S095029; Drug: pembrolizumab 200 mg (KEYTRUDA ®)

INTERVENTIONS:
Drug: S095029 — Participants will be treated with S095029 via intravenous (IV) infusion every 3 weeks (Q3W).
Drug: pembrolizumab 200 mg (KEYTRUDA ®) — Participants will be treated with 200 mg of pembrolizumab via intravenous (IV) infusion every 3 weeks (Q3W).

SUMMARY:
This study will investigate the safety, tolerability, and antitumor activity of S095029 (anti-NKG2A antibody) in combination with pembrolizumab in in microsatellite instability-high/Defective mismatch repair (MSI-H/dMMR) locally advanced unresectable or metastatic gastric /GEJ adenocarcinomas.

DETAILED DESCRIPTION:
This Phase 1b/2 study will be conducted in two parts; a safety lead-in part (Phase 1b) to identify the RP2D of S095029 in combination with pembrolizumab and an expansion part (Phase 2) to evaluate anti-tumor activity and safety in participants with locally advanced unresectable or metastatic MSI-H/dMMR gastric /GEJ adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of locally advanced and unresectable or metastatic gastric or gastro-esophageal junction adenocarcinoma
* Participants' tumor must have an MSI-H/dMMR status according to institutional guidelines and/or according to the College of American Pathologists, determined at any time prior to enrolment.

Exclusion Criteria:

* Has received more than one previous line of treatment in the locally advanced and unresectable or metastatic setting.
* Has received prior therapy with any checkpoint inhibitor (anti-PD-1, anti-programmed cell death ligand 1 (PDL1), anti-CTLA4).
* Participants who have received prior systemic anti-cancer therapy including investigational agents within 4 weeks (shorter interval, at least 5 half-lives, for kinase inhibitors or other short half-life drugs) prior to first study treatment.
* Prior radiotherapy if completed less than 2 weeks before first study treatment
* Major surgery less than 4 weeks prior to the first study treatment or participants who have not recovered from the side effects of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities (DLTs) | At the end of Cycle 1 (each cycle is 21 days)
  Phase 1b and Phase 2
Total Number of Adverse Events (AEs) | From screening to 90 days after the last dose
  Phase 1b and Phase 2
Adverse Events (AEs) Leading to Dose Interruption, Modification, or Delays | From screening to 90 days after the last dose
  Phase 1b and Phase 2
Adverse Events (AEs) Leading to Dose Discontinuation | From screening to 90 days after the last dose
  Phase 1b and Phase 2
Objective Response Rate (ORR) | Approximately 2 years
  Phase 2 ONLY. The Proportion of participants who achieve complete response (CR) or partial response (PR), as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Approximately 2 years
  Phase 1b and Phase 2. The time from the first documentation of complete response (CR) or partial response (PR) until the documented progressive disease (PD) or death, as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST).
Progression-Free Survival (PFS) | Approximately 2 years
  Phase 1b and Phase 2. The time from the first dose of S095029 to first documented PD or death due to any cause, whichever occurs first, as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST).
Disease Control Rate (DCR) | Approximately 2 years
  Phase 1b and Phase 2. The proportion of participants who achieved stable disease (SD), PR, or CR (based on participant's best response), as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST).
Overall Survival (OS) | Approximately 2 years
  Phase 1b and Phase 2. The time from first S095029 dose to death due to any cause.
Trough Concentrations of S095029 (Ctrough) | From first dose to 30 days after the last dose
  Phase 1b and Phase 2.
Concentration of potential antibodies directed against S095029 | From screening to 30 days after the last dose, or end of study if clinically indicated
  Phase 1b and Phase 2.
Objective Response Rate (ORR) | Approximately 2 years
  Phase 1b ONLY. The Proportion of participants who achieve complete response (CR) or partial response (PR), as per immune Response Evaluation Criteria in Solid Tumors (iRECIST).

CONTACTS AND LOCATIONS:
Locations (49):
- United States (3):
  - Ocala Oncology Center Pl, Ocala, Florida
  - Investigative Clinical Research of Indiana, Llc, Noblesville, Indiana
  - MD Anderson Cancer Center, Houston, Texas
- The Queen Elizabeth Hospital, Woodville South, Australia
- Austria (3):
  - Ordensklinikum Linz, Linz, Upper Austria
  - Med Universitat Wien-Allgemeines Krankenhaus Der Stadt Wien (AKH), Vienna, Vienna
  - Landeskrankenhaus (SALK), Salzburg
- Belgium (2):
  - UZ Leuven Campus Gasthuisberg, Leuven
  - Chu de Liege, Liège
- Brazil (5):
  - Cepon - Centro de Pesquisas Oncologicas, Florianópolis
  - Supera Oncologia, Santa Catarina
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Instituto Brasileiro de Controle Do Câncer, São Paulo
  - Hospital Albert Einstein, São Paulo
- Mount Sinai Hospital, Toronto, Canada
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital Institute, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine Qingchun Branch, Hangzhou, Zhengjiang Province
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Chru Lille - Hopital Claude Huriez, Lille
  - Institut Curie, Saint-Cloud
  - Inst. de Cancer de L'ouest, Saint-Herblain
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Bugat Pal Hospital, Gyöngyös
  - Bekes Megyei Kozponti Korhaz, Gyula
- Italy (5):
  - A.O.U. Seconda Università Degli Studi Di Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumor, Milan
  - A.O.U. Pisana-Ospedale Santa Chiara, Pisa
  - Policlinico Universitario Agostino Gemelli, Rome
  - Policlinico G.B. Rossi A.O.U.I. Di Verona, Verona
- Japan (3):
  - Cancer Institute Hospital of Jfcr, Koto-Ku, Tokyo
  - National Cancer Center Hospital, Chou-ku
  - Osaka International Cancer Institute, Osaka
- Pan American Center For Oncology Trials, Llc, Rio Piedras, Puerto Rico
- Spain (4):
  - University Hospital Vall D'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario de Valencia, Valencia
- United Kingdom (2):
  - The Royal Marsden in Chelsea, London
  - The Royal Marsden in Sutton, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/